CLINICAL TRIAL: NCT02972073
Title: Investigation of Trunk Neuromuscular Control in Patients With Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Peemongkon Wattananon, Principal investigator, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRG5880133
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain
Keywords: Low back pain; Neuromuscular control
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise intervention (Experimental): There are 4 different exercise interventions (4 independent intervention studies) based on different concepts in this entire project. Interventions include:
  1. core stabilization exercise
  2. movement system impairment approach
  3. neuromuscular activation using suspension
  4. kinematic linkage imbalance
  Interventions: Other: Exercise intervention
- Healthy control (No Intervention): This healthy control group will be informed to maintain usual daily activities and avoid participating in activities that involve trunk muscle exercise

INTERVENTIONS:
Other: Exercise intervention — Physical therapist will provide exercise for patients with low back pain for 60 minutes per day, 2-3 days per week for the total of 8 weeks.
  Arms: Exercise intervention

SUMMARY:
The purposes of this study include 1) determine clinical utility of clinical observation of aberrant movement patterns during functional trunk and pelvic movements in asymptomatic individuals and patients with non-specific low back pain, 2) characterize trunk neuromuscular control in asymptomatic individuals and patients with non-specific low back pain, and 3) determine the appropriate physical therapy intervention that addresses trunk neuromuscular control deficits in patients with non-specific low back pain.

DETAILED DESCRIPTION:
This study will use a sample of convenience between the ages of 21 - 65. Patients with non-specific low back pain (NSLBP) will be recruited by advertisement in 2 Mahidol university physical therapy clinics and participating clinics and hospitals. Asymptomatic participants will be also recruited by flyers posted in 2 Mahidol university physical therapy clinics.

Based upon power analysis for change in kinematic pattern in patients with NSLBP after an 8-week core stabilization exercise program, a total required sample size is 29 patients with NSLBP to detect a medium effect size (Cohen's d) of .48 at level (α) of .05 and power (1-β) of .80. Fifteen percent drop-out rate is used as a conservative sample size calculation. Therefore, 34 patients with NSLBP (29 X 15% drop-out) and 34 age-, sex-, and BMI-matched asymptomatic participants will be included for each independent intervention study (core stabilization exercise approach, movement system impairment approach, neuromuscular activation using suspension, and kinematic linkage imbalance approach). Each intervention will be separately collected and analyzed. The total of 272 participants will be recruited to fulfill this study project (4 independent intervention studies). However, sample size for asymptomatic participants can be decreased if participant from one intervention study is matched with patients with NSLBP in other intervention studies.

Patients with NSLBP who are interested in participation will undergo a screening process using inclusion-exclusion criteria checklist and receive brief information regarding the study. If they meet all inclusion criteria, the consent process and biomechanical testing will be scheduled. On date of consent and biomechanical testing, both asymptomatic participants and participants with NSLBP will be provided a consent form. To ensure they understand the study, they will be simply asked regarding the study (i.e. objectives, benefits, etc.) before signing the consent form. After the participants provide a written informed consent, they will undergo a standardized physical therapy examination performed by an experienced physical therapist (PT-A). For patients with NSLBP, they will also complete 3 clinical outcome measures including 1) numeric pain rating scale (Thai version), 2) Oswestry disability index (Thai version), and 3) general health status questionnaire (Thai version). This pre-biomechanical data collection process will last approximately 60 minutes.

For biomechanical testing, body landmarks will be identified and marked with a skin pen for 4 motion sensors and 16 pairs of surface electromyography (EMG) electrodes in lower back and abdominal areas. Any hair in the area around the sensors and electrodes will be shaved. Before placing surface EMG electrodes, the skin will be lightly abraded using abrasive paper and cleaned using cotton with alcohol to lower the skin impedance. Electrodes will be aligned parallel to the muscle fibers. This process will take approximately 30 minutes. Then, participants will proceed to the biomechanical testing which includes 1) trunk muscle strength test, 2) functional trunk and pelvic movement tests, and 3) core control tasks.

Trunk muscle strength test Strength test Participants will wear a climbing harness connecting with a tension load cell and sit in a testing apparatus in a neutral trunk position with pelvic securely locked. This apparatus intends to reduce compensation from lower extremities during sub-maximal (15% of body weight) and maximal voluntary isometric contractions. Participants will be instructed to use their trunk gradually pulling the load cell (isometric contraction in neutral trunk position) for 10 seconds in forward, backward, and 2 side bending directions. Participants will be given 2 practice trials in each direction to adjust the force and reduce a learning effect. Visual feedback of force to sub-maximal target will be provided. Two trials of sub-maximal voluntary isometric contractions will be collected in each direction. Only 1 trial of maximal voluntary isometric contraction will be collected to avoid muscle fatigue (in both asymptomatic participants and patients with NSLBP) and pain exacerbation (in patients with NSLBP). The intention of collecting maximal contraction data is to use for EMG standardization. Participants will rest in between each trial to minimize fatigue. Pain and rating perceived exertion (RPE) will be monitored and recorded at the end of trunk strength test. This protocol will take approximately 15 minutes.

Functional trunk and pelvic movement tests Participants will stand on a drawing paper with feet shoulder width apart in front of the motion transmitter. The foot print will be drawn using a marker. This foot print will be used for post-test positioning. The participants will stand in a natural stance facing away from the transmitter with arms down by sides. Participants will be instructed to stand up straight and maintain that position for digitization. After the completion of digitization, participants will be instructed to perform functional movements including 1) active forward bend and return to upright position, 2) right and left straight leg raise tests, 3) right and left hip abduction with knee flexion tests, 4) quadruped backward rock test, 5) prone with right and left knee flexion tests, 6) prone with right and left hip internal/external rotation tests, and 7) prone with right and left hip extension tests. Participants will perform 2 trials of 3 consecutive repetitions of each functional movement tests. Two physical therapists (PT-B and PT-C), who are blinded to the group membership, will simultaneously observe and independently rate aberrant movement patterns during biomechanical data collection. This protocol will take approximately 30 minutes.

Core control tasks Participants will sit on an unstable chair with feet supported. The chair is mounted on a half ball that makes the chair unstable and tilt. Participants will be instructed to balance the chair without tipping the chair in any direction. The participants will maintain upright seated balance with crossing both arms in front of their chest. The participants will have an opportunity to get familiar with the balance testing protocol prior to the data collection to minimize the learning effect. This core control tasks aim to investigate the performances that represent static and dynamic stabilities of the trunk. For static stability, the participants will perform 3 trials of 60-second seated balance tests with their eyes open, and 3 trials of 60-second seated balance tests with their eyes closed. The participants will be given a 1-minute rest period between trials to avoid muscle fatigue. For dynamic stability, the participants will be instructed to perform a dynamic stability using lumbar spine (without trunk leaning to tilt an unstable chair as far as they can) in 8 different directions (forward, backward, right, left, right diagonal, and left diagonal). The participants will be given 1 practice trial to reduce possibility of learning effect, and 3 real trials with 1-minute rest period between trials. Pain and RPE will be recorded at the completion of core control task. This protocol will take approximately 30 minutes.

Patients with NSLBP will be assigned to one of different physical therapy interventions according to participating clinics and hospitals, while asymptomatic participants will be encouraged to maintain usual daily activities and avoid participating in activities that involve trunk muscle exercise. After completion of an 8-week physical therapy intervention, both asymptomatic participants and patients with NSLBP will undergo the standardized physical therapy examination and biomechanical data collection again. For patients with NSLBP, they will also complete clinical outcome measures for post physical therapy intervention.

Physical therapy intervention Patients with NSLBP will be treated with a standard physical therapy intervention based upon different treatment concepts. In general, these interventions include strengthening exercise, endurance exercise, stretching exercise, patient education, patient ergonomics, and home exercise program. There is no reported adverse effect of those physical therapy interventions. Therefore, those physical therapy interventions are safe for treating patients with NSLBP. Each patient will be treated 1-2 times per week for 60 minutes each session for 8 weeks by experienced physical therapists. Patients will be given a home exercise log for exercise compliance.

All Statistical analyses will be performed using statistical package for the social science (SPSS) software (IBM SPSS Statistics for Windows, Version 21.0., New York, USA).

Study objective 1 is to determine inter-rater reliability and diagnostic accuracy of clinical observation of aberrant movement patterns during functional trunk and pelvic movements in patients with NSLBP. Agreement on the presence/absence of aberrant movement patterns between physical therapists (PT-B and PT-C) will be determined using separate kappa statistics. Diagnostic accuracy will be determined using accuracy statistics which include sensitivity, specificity, and likelihood ratio. Significance level will be held at .05 for all analysis. Confidence intervals will also be calculated.

Study objective 2 is to characterize neuromuscular control in asymptomatic participants and patients with NSLBP during functional activities. Each variable will be analyzed separately. Descriptive statistics (i.e. mean and standard deviation) will be performed and statistical assumptions (i.e. normal distribution, homogeneity of variance, etc.) related to specific statistical tests will be performed. Statistical transformation will be performed if appropriate. Then, statistical test (i.e. independent t-test, Mann-Whitney U-test, etc.) that appropriate to the data will be performed to determine the difference between asymptomatic participants and patients with NSLBP. Significance level will be held at .05 for all analyses. Post-hoc power analysis will also be performed to determine statistical power and effect size.

Study objective 3 is to determine the appropriate physical therapy intervention that addresses neuromuscular control deficits in patients with NSLBP. First, the effects of each physical therapy intervention on trunk neuromuscular control and clinical outcomes will be determined. Prior to utilization of statistical tests, descriptive statistics will be performed and statistical assumptions will be tested. Transformation will be performed if the data are not normally distributed. Appropriate statistical tests will be performed to determine the effects of each physical therapy intervention on neuromuscular control and clinical outcome. Significance level will be held at .05 for all analyses. Post-hoc power analysis will be performed. In addition, this study objective will determine the ability of physical therapy intervention on matched- and unmatched-intervention patients based upon each intervention criteria. Each patient with NSLBP will be classified based upon clinical criteria of each physical therapy intervention. Pre-post difference for matched and unmatched groups will be compared using appropriate statistical tests. Significance level will be held at .05 for all analyses. Post-hoc power analysis will also be performed.

ELIGIBILITY:
Inclusion Criteria for patients with non-specific low back pain:

* Between the ages of 21 and 65
* Current episode of back pain less than 3 months which they seek medical intervention
* Numeric pain rating scale (NPRS) greater than 5 on an 11-point scale (0 = no pain, 10 = worst pain ever)
* Oswestry disability score (Thai version) greater than 50%
* No medical or professional health care intervention including physical therapy for low back pain in last 6 months

Inclusion Criteria for healthy individual:

* Between the ages of 21 and 65
* No episode of back pain for 3 months prior to the participation
* No regular exercise routine that is composed of core stabilization exercise.

Exclusion Criteria for both groups:

* Clinical signs of systemic disease
* Definitive neurologic signs including weakness or numbness in the lower extremity
* Previous spinal surgery
* Diagnosed osteoporosis, severe spinal stenosis, and/or inflammatory joint disease
* Pregnancy
* Any lower extremity condition that would potentially alter trunk movement in standing
* Vestibular dysfunction
* Extreme psychosocial involvement
* Body mass index (BMI) greater than 30 kg/m2
* Active treatment of another medical illness that would preclude participation in any aspect of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) muscle activity | Change from baseline muscle activity at 8 weeks after exercise intervention.
  Muscle activity recorded by surface-electromyography (EMG) during functional movements will be used to determine muscle activation pattern changes at 8 weeks after exercise intervention.
Kinematic pattern of movement | Change from baseline movement pattern at 8 weeks after exercise intervention.
  Patterns of functional movement will be captured using electromagnetic tracking system and used to determine changes in kinematic pattern of movement at 8 weeks after exercise the exercise intervention.

SECONDARY OUTCOMES:
Numeric pain rating scale | Change in pain from baseline at 8 weeks after exercise intervention
  Pain assessed by a numeric pain rating scale will be used to determine change in pain at 8 weeks after exercise intervention.
Oswestry disability index | Change from baseline disability level at 8 weeks after exercise intervention
  Disability level measured by Oswestry disability index will be used to determine change in disability level at 8 weeks after exercise intervention.
Short-form general heath status (SF-36) questionnaire | Change from baseline general health status at 8 weeks after exercise intervention
  General health status assessed by short-form general health status questionnaire (SF-36) will be used to change in general health status at 8 weeks after exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No
Only demographic and clinical outcome data will be made available for other researchers upon request after the end of the study

REFERENCES:
- [Background] Biely SA, Silfies SP, Smith SS, Hicks GE. Clinical observation of standing trunk movements: what do the aberrant movement patterns tell us? J Orthop Sports Phys Ther. 2014 Apr;44(4):262-72. doi: 10.2519/jospt.2014.4988. Epub 2014 Jan 22. PMID 24450372
- [Background] Hicks GE, Fritz JM, Delitto A, McGill SM. Preliminary development of a clinical prediction rule for determining which patients with low back pain will respond to a stabilization exercise program. Arch Phys Med Rehabil. 2005 Sep;86(9):1753-62. doi: 10.1016/j.apmr.2005.03.033. PMID 16181938
- [Background] Spinelli BA, Wattananon P, Silfies S, Talaty M, Ebaugh D. Using kinematics and a dynamical systems approach to enhance understanding of clinically observed aberrant movement patterns. Man Ther. 2015 Feb;20(1):221-6. doi: 10.1016/j.math.2014.07.012. Epub 2014 Jul 24. PMID 25116648